CLINICAL TRIAL: NCT07146685
Title: Effect of Local Anesthetic Concentration on Rebound Pain: A Randomized Control Study
Acronym: RPRCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Leon Grinman, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 302714
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Rebound Pain; Shoulder Arthroplasty; Interscalene Block
Keywords: local anesthetics; rebound pain; brachial plexus; shoulder arthroscopy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized control study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concentrated (Active Comparator): Standard management of higher percent local anesthetic: 0.5% Bupivacaine
  Interventions: Drug: Bupivacaine
- Dilute (Experimental): More dilute local : 0.25% Bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — We are comparing two concentrations of the same drug: 10 ml of 0.5% and 20 ml of 0.25%; We will use the same milligram dose (50 mg).

SUMMARY:
Randomized control study that compares different concentrations of local anesthetic to investigate whether a lower concentration of local anesthetic would contribute to lower rebound pain scores at 24 hours post op in patients undergoing anatomic or reverse total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Total shoulder replacement patients (anatomic and reverse)
* Adult patients (greater than or equal to 18 years)
* Any gender
* Any race

Exclusion Criteria:

* - Chronic Pain diagnoses including:
* substance/opioid use disorder
* complex regional pain syndromes
* fibromyalgia
* Daily persistent opioid use spanning 3 months prior to surgery date
* Allergy to local anesthetics or NSAIDS
* Respiratory pathologies including:
* CPAP- non-compliant / untreated obstructive sleep apnea
* COPD
* Restrictive lung disease (pulmonary fibrosis, interstitial pneumonia, etc)
* Contralateral diaphragm dysfunction
* BMI > 40
* Ipsilateral extremity pre-existing nerve injury
* GFR < 60
* NSAID contraindications
* Inability to follow up
* Revision surgery
* Patients requesting block as primary (avoidance of general anesthesia)
* Need or request for brachial plexus catheter or liposomal bupivacaine
* Vulnerable populations (pregnancy, incarceration, etc)
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Max NRS Pain Score at 24 hours | 24 hours after intervention; will also be assessed at 48 and 72 hours, though these are not the primary outcome for the study.
  Patients will be Assessed 24 hours after intervention for a pain score between 0 and 10, 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Qor15 score questionnaire. | 24, 48 and 72 hours.
  Patient will answer QoR15 questionnaire
Lowest NRS pain score | 24, 48, 72 hours
  Patient will be assessed for lowest NRS pain scores
Opioid Use | Assessed at 72 hours
  Total doses used will be converted to MMEs.
Sensory Block Duration | Assessed at 24 hours.
  We will ask the patient how long they felt the nerve block was effective, in terms of hours.
Presence of dyspnea/shortness of breath | Assessed at 24 hours.
  We will ask the patient if they ever had trouble breathing or shortness of breath during the duration of the block.
Presence of Nausea or Vomiting | 24, 48, 72 hours
  We will ask the patient if there was any incidence of nausea or vomiting.
Presence of persistent paresthesia | 24, 48, and 72 hours.
  We will ask the patient if there is any presence of persistent paresthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Leon N Grinman, DO, Principal Investigator — UVA
Locations (1):
- UVA Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
The details of the IPD Plan are unknown at this time, but it will likely be shared.

REFERENCES:
- [Background] Al-Kaisy A, McGuire G, Chan VW, Bruin G, Peng P, Miniaci A, Perlas A. Analgesic effect of interscalene block using low-dose bupivacaine for outpatient arthroscopic shoulder surgery. Reg Anesth Pain Med. 1998 Sep-Oct;23(5):469-73. PMID 9773699
- [Background] Fredrickson MJ, Abeysekera A, White R. Randomized study of the effect of local anesthetic volume and concentration on the duration of peripheral nerve blockade. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):495-501. doi: 10.1097/AAP.0b013e3182580fd0. PMID 22664978
- [Background] Lee HJ, Woo JH, Chae JS, Kim YJ, Shin SJ. Intravenous Versus Perineural Dexamethasone for Reducing Rebound Pain After Interscalene Brachial Plexus Block: A Randomized Controlled Trial. J Korean Med Sci. 2023 Jun 19;38(24):e183. doi: 10.3346/jkms.2023.38.e183. PMID 37337808
- [Background] Woo JH, Lee HJ, Oh HW, Lee JW, Baik HJ, Kim YJ. Perineural dexamethasone reduces rebound pain after ropivacaine single injection interscalene block for arthroscopic shoulder surgery: a randomized controlled trial. Reg Anesth Pain Med. 2021 Nov;46(11):965-970. doi: 10.1136/rapm-2021-102795. Epub 2021 Sep 17. PMID 34535548
- [Background] Uppal V, Barry G, Ke JXC, Kwofie MK, Trenholm A, Khan M, Shephard A, Retter S, Shanthanna H. Reducing rebound pain severity after arthroscopic shoulder surgery under general anesthesia and interscalene block: a two-centre randomized controlled trial of pre-emptive opioid treatment compared with placebo. Can J Anaesth. 2024 Jun;71(6):773-783. doi: 10.1007/s12630-023-02594-0. Epub 2023 Oct 13. PMID 37833472
- [Background] Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth. 2021 Apr;126(4):862-871. doi: 10.1016/j.bja.2020.10.035. Epub 2020 Dec 31. PMID 33390261
- [Background] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Background] Lavand'homme P. Rebound pain after regional anesthesia in the ambulatory patient. Curr Opin Anaesthesiol. 2018 Dec;31(6):679-684. doi: 10.1097/ACO.0000000000000651. PMID 30124544